CLINICAL TRIAL: NCT05908006
Title: Comparison of Steatosis and Fibrosis Measurements From Velacur and MRE/MRI-PDFF in Patients With Chronic Liver Disease
Brief Title: Validation Study of the Velacur System in Comparison to MRE & MRI-PDFF in Patients With (Suspected) Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: GI Alliance (Other)
Collaborators: Sonic Incytes (Industry)
Responsible Party: Sponsor
Other Study IDs: Velacur-2
Record Dates: First submitted 2023-03-29; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Non-alcoholic Fatty Liver Disease (NAFLD)
Keywords: NASH; NAFL
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- non-randomized, open-label study: All participants will have the same Laboratory and Diagnostic Assessments and Imaging Procedures.
  Interventions: Device: Velacur

INTERVENTIONS:
Device: Velacur — Imaging Procedures Comparison
  Other Names: MRE/MRI; Fibroscan

SUMMARY:
The goal of this open-label, non-randomized, prospective study is to compare Velacur and MRE in all sexes, 18-80 years old with Non-Alcoholic Fatty Liver Disease (NAFLD). The main aims is to:

* Validate the use of Velacur and elastography cut offs in a patient cohort with all types of chronic liver disease, against MRE results for fibrosis staging.
* Validate the use of Velacur and attenuation cut offs in a patient cohort with all types of chronic liver disease, against MRI-PDFF results for steatosis staging.

Participants will Study participants will attend 1 study visit, in which measurement of liver stiffness with Velacur and FibroScan, will be performed by a certified technician. As part of Visit 1, Patients will also complete an MRI exam which will include both MRE and MRI-PDFF measurements (MRI imaging can take place within 28 days of the Velacur scan).

DETAILED DESCRIPTION:
This will be a prospective, open label, validation study of the Velacur system in comparison to MRE and MRI-PDFF in patients with liver disease or suspected liver disease.

Approximately 100 subjects may be enrolled in this study. Participants should span all levels of fibrosis and steatosis.

The study is comprised of: Screening Period (up to 8 days) and Visit 1. There are no safety follow-up visits in this study.

The primary objective of the study is to compare the results of Velacur against MRE and MRI-PDFF results for liver stiffness and steatosis. As part of prior studies, using MRE as the gold standard, clinical cut-off for Velacur have been developed. The primary objective of this study is to validate these cut-offs to see if Velacur can correctly classify patients.

Secondary objectives include correlating the stiffness and attenuation results of Velacur with other clinical measures of fibrosis and steatosis such as Fib-4, and correlations with other clinical measurements collected through clinical care or clinical trials, such as Enhance Liver Fibrosis (ELF) test, FibroScan, MRI, or ultrasound based shear wave elastography (SWE) as they are available.

ELIGIBILITY:
Inclusion Criteria:

Patients with evidence of NAFLD or other chronic liver disease such as one of the following:

Biopsy proven chronic liver disease OR

Evidence of hepatic steatosis or chronic liver disease on non-invasive assessment by one or more of the following criteria:

* Abdominal ultrasound within 12 months
* MRI-PDFF (greater than 12%) within 12 months
* FibroScan CAP score > 230 dB/m within 12 months OR At least 2 criteria for metabolic syndrome and increased stiffness on FibroScan (>8kPa) within 12 months

Exclusion Criteria:

* BMI greater than 40 kg/m2 (or unable to fit into MRI bore)
* Subject with current, significant alcohol consumption or history of significant alcohol consumption
* Subjects with evidence of decompensated liver disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All sexes, 18-80 years old. Patients with Non-Alcoholic Fatty Liver Disease (NAFLD), including both those with Non-Alcoholic Fatty Liver (NAFL) and Non-Alcoholic Steatohepatitis (NASH).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-07-15 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Elasticity measurements | 2024
  Validate the use of Velacur and elastography cut offs with all types of chronic liver disease, against MRE results for fibrosis staging. The liver tissue elasticity is measured in kilopascals (kPa), using Velacur.
  The Velacur elasticity measurements will be compared to those from Magnetic Resonance Elastography, which is measuring liver tissue elasticity in kilopascals (kPa).
Attenuation measurement | 2024
  Validate the use of Velacur and attenuation cut offs with all types of chronic liver disease, against MRI-PDFF results for steatosis staging. Ultrasound attenuation is a quantitative measurement of ultrasound image parameters. Attenuation is measured by Velacur, and uses units of of decibels per meter (dB/m).
  These numbers are compared to the fat percentage as measured by MRI proton density fat fraction, which is measured in percentage fat (%).

SECONDARY OUTCOMES:
Serum markers such as Fib-4, APRI and NALFD Fibrosis score or ELF (enhanced liver fibrosis) score. | 2024
  Comparison of Velacur stiffness and attenuation results with other clinical measures of fibrosis and steatosis, such as blood work, using readily available scores and attenuation results with other clinical measures of fibrosis and steatosis, such as blood work, using readily available scores.
The combined outputs of elasticity and attenuation from Velacur and FibroScan | 2024
  Discriminatory ability of Velacur compared with other noninvasive markers, such as FibroScan

OTHER OUTCOMES:
Elasticity and attenuation measurements from the Velacur system and BMI measurements (kg/m2) | 2024
  Evaluate Velacur to measure liver stiffness and attenuation in patients of varying body composition
Comparison of previously calculated cutoff, with new measurements. | 2024
  Evaluate the cutoffs based on this cohort of patients, in comparison to previous cutoffs

CONTACTS AND LOCATIONS:
Overall Officials: Sri Naveen Surapaneni, MD, Principal Investigator — GI Alliance; Reed B Hogan, III, MD, Principal Investigator — GI Alliance
Locations (2):
- United States (2):
  - GI Alliance-Flowood, MS, Flowood, Mississippi
  - GI Alliance-Webster, TX, Webster, Texas